CLINICAL TRIAL: NCT05890625
Title: The Effect of the Responsive Web-based Roadmap (InT-mAp) in Infertility Treatment on Women's Drug Administration, Treatment Success and Anxiety.
Brief Title: Responsive Web-based Roadmap (InT-mAp) in Infertility Treatment
Acronym: InT-mAp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maltepe University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Tuğba Bozdemir, Lecturer, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022/20-02
Record Dates: First submitted 2023-05-18; First posted 2023-06-06 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Infertility, Female; Web; Anxiety; IVF
Keywords: infertility; web-based education; drug administration; treatment success; anxiety
MeSH Terms: conditions — Infertility, Female; Anxiety Disorders; Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- InT-mAp (Experimental)
  Interventions: Other: InT-mAp
- Control group (Active Comparator)
  Interventions: Other: On going treatment

INTERVENTIONS:
Other: On going treatment — No additional attempts will be made by the investigator on the cases in the control group. These cases will only benefit from the services in the clinic.
  Arms: Control group
Other: InT-mAp — InT-mAp, the content of which will be created as a result of the evaluation of the nursing needs of infertile women, consists of a web-based training and online consultancy platform. The treatment plan specific to each participant will be entered into the web base individually, and the participants will be able to follow and manage the treatment protocols and appointments under their own control. InT-mAp is a guide that helps breakers about the intended use, effects, side effects of the drugs under treatment and how to self-administer, especially for women.
  Arms: InT-mAp

SUMMARY:
Infertility affects approximately 48 million couples and 186 million individuals globally, and it has biological, psychosocial, and economic problems in couples. It is a vital global reproductive health problem that has burdens and affects not only families but also society and the state.

Studies indicate that many situations experienced during the infertility treatment process negatively affect the treatment results, and the anxiety of individuals receiving treatment, especially women, is high. The previous literature reports that during the infertility treatment process, women experience a decrease in their anxiety and self-confidence about drug administration, they have doubts about the dose, administration, and time of drugs, and the rate of mistakes made regarding drug administration is too high to be ignored. Such cases may lead to cycle cancellations in infertility treatment, interrupting the treatment, adversely affecting the success of the treatment, and thus exposing the couple to more than one treatment trial. The interruption of the treatment with the cycle cancellation, the increase in the number of treatment attempts, the repetitions cause the woman to be exposed to a higher amount of drug, the cost to increase with each treatment trial, an increase in the economic burden of the couples, and an increase in the financial burden for the country. In addition to these physical and economic burdens, feelings such as anxiety, concern, hopelessness, and depression increase in couples, and they may eventually experience burnout.

In order to improve the care of infertile individuals, it is clearly stated in the literature that couples need open communication channels with health care professionals, obtaining qualified information, instilling realistic hope, empowerment, accessibility of care services, and they have unmet and high-quality care needs. The increase in the use and use of web-based education services in the globalizing world gives us hope in providing a solution to this issue.

This project was mainly designed to answer the question of "Is the responsive web-based roadmap (InT-mAp) developed in solving the problems encountered in drug administration, treatment success and reducing anxiety in infertile women treated with Assisted Reproductive Techniques (ART)?"

With InT-mAp, which investigators will develop using web-based education technology, which is a distance education method in this age of technology; investigators aimed to reduce/reduce the margin of error in ART treatment-drug practices, to contribute positively to the treatment process, and to reduce the social, economic and psychological burdens by reducing the anxiety level of individuals in this process. Besides, the InT-mAp, which will be developed to meet individuals' education and counseling needs for general infertility issues and the treatment process, will reduce the workload of healthcare professionals working in this field and make a positive contribution to drug administration consultancy.

With this study, investigators aimed to provide participants with time-saving, individualized care, to reach the right information whenever they want, regardless of time and place, on every subject they need in the field of infertility. Investigators predict that sufficient follicle development, healthy oocytes and pregnancy can be achieved by creating awareness in infertile women and minimizing the conditions that may adversely affect the treatment process and results. Contributing to the health and economic indicators of the country by reducing cycle cancellations and reducing costs are among our important goals. The most important features that make the project unique are the absence of online support and a sensitive web-based training platform, where the infertility treatment process in Turkey can be followed in detail by the users, and individualized care and training needs are met.

ELIGIBILITY:
Inclusion Criteria:

* In vitro fertilization-Embryo transfer (IVF-ET)/ Intracytoplasmic Sperm Injection (ICSI)-ET treatment planned as assisted reproduction treatment (ART) and who are in the controlled ovarian hyperstimulation (COS) process of the treatment,
* Having no psychological or chronic illness and related treatment that may affect the success of treatment other than the cause of infertility,
* Primary infertile,
* Being under 35 years old,
* Able to speak, read and write Turkish, perceive and answer questions correctly and communicate effectively,
* Having a smart phone with Android and the operating system for i-Phone (IOS) operating systems, being able to use mobile applications, and having sufficient equipment to use these applications (internet, etc.),
* Women who volunteered to participate in the study will be included in the sample.

Exclusion Criteria:

* Not meeting the sampling criteria,
* Wanting to leave after the start of work,
* Women with errors or deficiencies in their evaluation/use of the mobile application will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change from Anxiety Level at 12 weeks | It will be administered before controlled ovarian hyperstimulation treatment and after embryo transfer. (At 0 and approx. at 12 weeks))
  Beck Anxiety Inventory: The minimum score to be taken from the scale is 0, and the maximum score is 63.
Pregnancy rate | 12 days after embryo transfer (approx. at 13 weeks)
  Human chorionic gonadotropin (B-hCg)
Treatment success | After controlled ovarian hyperstimulation treatment (at 4 weeks)
  Follicle count (Number of follicles formed after controlled ovarian hyperstimulation)
Treatment success | After controlled ovarian hyperstimulation treatment (at 4 weeks)
  Oocyte count (Number of oocytes formed after controlled ovarian hyperstimulation)(
Cycle success | After controlled ovarian hyperstimulation treatment (approx. at 12 weeks)
  Embryo transfer rate (embryo transfer status)
Nursing Needs of Infertile Women | before the treatment (at 0 week)
  Nursing Needs Assessment Scale For Women With Infertility: The lowest score that can be obtained from the scale is 18, and the highest score is 72.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Zeynep Kamil Kadın ve Çocuk Hastalıkları Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No